CLINICAL TRIAL: NCT07226518
Title: Robot-assisted Gait Training and Transcutaneous Spinal Cord Stimulation in Chronic Non-ambulatory Stroke Survivors: Pilot RCT Trial
Brief Title: Walking and tSCS in Non-ambulatory Stroke Survivors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Wen Liu, Ph.D., Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STUDY00162114
Record Dates: First submitted 2025-11-04; First posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Chronic Stroke Survivors; Chronic Stroke Patients; Stroke
Keywords: stroke gait rehabilitation; Transcutaneous spinal cord stimulation; Non invasive spinal cord stimulation; Robot assisted gait training
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Robot assisted gait training combined with Transcutaneous spinal cord stimulation (Experimental)
  Interventions: Device: Robot-assisted gait training and transcutaneous spinal cord stimulation in chronic non-ambulatory stroke survivors: pilot RCT trial
- Robot assisted gait training alone (Active Comparator)
  Interventions: Device: Robot assisted gait training alone

INTERVENTIONS:
Device: Robot-assisted gait training and transcutaneous spinal cord stimulation in chronic non-ambulatory stroke survivors: pilot RCT trial — Participants in the experimental group will receive 30 minutes of robot assisted gait training (RAGT) transcutaneous spinal cord stimulation 3 times per week, 8 weeks, totaling 24 sessions. The gait training will utilize a treadmill equipped with a partial-body-weight support system and a lab-developed RAGT device. The RAGT protocol will be the same as in the control group
  Arms: Robot assisted gait training combined with Transcutaneous spinal cord stimulation
Device: Robot assisted gait training alone — Participants in the control group will receive 30 minutes of assisted gait training (RAGT), 3 times per week, for 8 weeks, totaling 24 sessions. The gait training will utilize a treadmill equipped with a partial-body-weight support system and a lab-developed RAGT device
  Arms: Robot assisted gait training alone

SUMMARY:
Rehabilitation interventions commonly used for stroke survivors include task-specific training, balance and strength exercises, and the use of assistive devices to enhance mobility and independence. Advanced technologies, such as body-weight-supported treadmill systems and robotic devices, may be employed when appropriate. Current rehabilitation therapies for stroke survivors are moderately effective with a limited effect size, especially in stroke survivors with severe impairment. Novel therapies, such as transcutaneous spinal cord stimulation (tSCS), may further improve outcomes in the target population. This pilot study will allow us to examine the feasibility and gather pilot data on a combined intervention of assistive gait training and tSCS in non-ambulatory stroke survivors.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years at time of consent
2. All genders included.
3. Chronic ischemic or hemorrhagic stroke >=6 months, with limited within-home comfortable walking speed <= 0.49 m/s and unable to walk independently in community (FAC <= 3)
4. Able to communicate with investigators, follow 2-step command, and correctly answer consent comprehension questions in English.
5. Currently not participating in treadmill walking exercises or exercises involving weight-bearing activities.
6. Have physicians' approval for exercise and be in a stable medical condition

Exclusion Criteria:

1. Hospitalization for cardiac or pulmonary disease within the past 3 months
2. Have musculoskeletal disorders that prevent the participant from participating in the exercise
3. Blood pressure higher than 200/110 mm Hg
4. Significant ataxia or unilateral spatial neglect (score of 2 on NIH stroke scale item 7 or 11)
5. Reported pain that limits or interferes with activities of daily living and physical activity/exercise
6. Diagnosis of other neurological diseases (multiple sclerosis, Alzheimer's disease, Parkinson's disease)
7. Diagnosis of severe depression (HADS score 15-21)
8. Unable to speak or understand English, and travel to the research laboratory.
9. Contraindications to tSCS and TMS

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiac Output (Measured by Impedance Cardiography - BIOPAC MP160 System) | Before and after 24 training sessions (8 weeks)
  Cardiac output (L/min) will be measured using an impedance cardiography system (MP160, BIOPAC Systems Inc., Goleta, California). Measurements will be done during a 6-minute walk test. Data collection for each participant will occur at approximately the same time of day (between 9:00 AM and 11:00 AM) before the first intervention session and after completion of the 24th intervention session.

CONTACTS AND LOCATIONS:
Overall Officials: Wen Liu, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- Neuromuscular Research Laboratory, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided